CLINICAL TRIAL: NCT06954324
Title: Investigation of the Effect of Erector Spinae Plane Block on Systemic Immuno-Inflammatory Index in Breast Cancer Surgery: A Prospective Randomized Controlled Study
Brief Title: Investigation of the Effect of Erector Spinae Plane Block on Systemic Immuno-Inflammatory Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ahmet Gültekin, Associate Professor, Namik Kemal University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: NamikKU-AGultekin-Ezgi2025
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Erector Spinae Plane Block; Systemic Immune-inflammatory Index; Breast Cancer
Keywords: Breast cancer; Systemic immune inflammatory index (SII); Erector spinae plane block (ESPB); Stress response
MeSH Terms: conditions — Breast Neoplasms; Fractures, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental): Preoperative thoracic level 4 ESP block was applied
  Interventions: Procedure: Erector spinae plane block
- Control (No Intervention): Group with analgesia provided by Contromal (IM) without blockade

INTERVENTIONS:
Procedure: Erector spinae plane block — This study aims to compare the effects of erector spinae plane block (ESPB) and systemic tramadol use as postoperative analgesia methods on the systemic immune-inflammatory index (SII) in patients undergoing breast cancer surgery.
  Arms: Erector spinae plane block

SUMMARY:
Erector spinae plane block (ESPB) is a novel interfascial block technique first described by Forero in 2016. It has been reported to be effective in various clinical indications. In ESPB, local anesthetic is injected between the deep fascia of the erector spinae muscle and the transverse process of the vertebra, allowing cephalocaudal spread along the erector spinae muscle. The goal of the injection is to provide sensory blockade by affecting the anterior rami of the spinal nerves in the region.

ESPB has been used during breast and axillary lymph node surgeries to manage postoperative pain. In addition to tumor cells, immune and inflammatory cells such as neutrophils, platelets, and lymphocytes contribute to the dissemination and invasion of tumor cells into the peripheral circulation. Noninvasive biomarkers such as serum inflammatory markers are increasingly valued for their simplicity and predictive potential. Platelets have been shown to facilitate epithelial-mesenchymal transition of tumor cells; neutrophils support tumor adhesion via growth factors such as VEGF and proteases; lymphocytes play a role in modulating the host immune response to malignancy.

The systemic immune-inflammatory index (SII), calculated as (platelet count × neutrophil count) / lymphocyte count, is a relatively new composite marker that reflects immune and inflammatory responses. It has been evaluated as a prognostic biomarker in several cancer-related studies.

Postoperative pain and surgical stress activate systemic inflammatory responses. ESPB is performed as part of postoperative analgesia in patients undergoing breast cancer surgery under general anesthesia, based on voluntary participation. The aim of this study is to evaluate the effect of ESPB on postoperative SII levels in comparison to other analgesia modalities.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-75 years
* ASA (American Society of Anesthesiologists) physical status I-II-III
* Undergoing unilateral breast cancer surgery under general anesthesia
* Volunteered to participate in the study and signed informed consent

Exclusion Criteria:

* Allergy or contraindication to local anesthetics
* Coagulopathy or on anticoagulant therapy
* Infection at the injection site
* History of chronic pain or opioid use
* Neurological or psychiatric disorders affecting pain perception
* Refusal to receive regional anesthesia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female (because it is a breast cancer study)
Enrollment: 120 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Systemic Immune-Inflammation Index (SII) | 6 hours postoperatively
  Systemic immune-inflammation index (SII) will be calculated using the formula:
  SII = (Platelet count × Neutrophil count) / Lymphocyte count. This index will be used to evaluate the effect of erector spinae plane block (ESPB) on postoperative systemic inflammation in patients undergoing breast cancer surgery.

SECONDARY OUTCOMES:
Postoperative Pain Score | At 0, 2, 4, and 6 hours postoperatively
  Postoperative pain will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). Pain scores will be recorded at rest and during movement at predefined time points to evaluate the analgesic effectiveness of erector spinae plane block (ESPB).

CONTACTS AND LOCATIONS:
Locations (1):
- Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to privacy and confidentiality concerns, individual participant data (IPD) will not be made available to other researchers. The data will remain confidential, in accordance with institutional and regulatory guidelines.

REFERENCES:
- [Background] He W, Wu Z, Zu L, Sun H, Yang X. Application of erector spinae plane block guided by ultrasound for postoperative analgesia in breast cancer surgery: A randomized controlled trial. Cancer Commun (Lond). 2020 Mar;40(2-3):122-125. doi: 10.1002/cac2.12013. Epub 2020 Mar 16. No abstract available. PMID 32175686
- [Background] Liu J, Shi Z, Bai Y, Liu L, Cheng K. Prognostic significance of systemic immune-inflammation index in triple-negative breast cancer. Cancer Manag Res. 2019 May 14;11:4471-4480. doi: 10.2147/CMAR.S197623. eCollection 2019. PMID 31191009
- [Derived] Gulay E, Gultekin A, Yildirim I, Arar C, Ozkan Gurdal S. Comparison of erector spinae plane block and tramadol on postoperative systemic immune-inflammatory response in breast cancer surgery: A prospective randomized controlled trial. Medicine (Baltimore). 2025 Sep 12;104(37):e44466. doi: 10.1097/MD.0000000000044466. PMID 40958235